CLINICAL TRIAL: NCT07112456
Title: Nebulized Ketamine Plus Standard Care vs. Standard Care Alone in Moderate to Severe Asthma Exacerbations: A Randomized Clinical Trial (KET-AIR Trial)
Brief Title: Nebulized Ketamine Plus Standard Care vs. Standard Care Alone in Moderate to Severe Asthma Exacerbations
Acronym: KET-AIR
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oman Medical Speciality Board (Other Government)
Responsible Party: Principal Investigator, Al Mahanad Al Julandani, Emergency Medicine Resident Doctor, Oman Medical Speciality Board
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OMSB24030
Record Dates: First submitted 2025-07-22; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Asthma Acute; Asthma Attack; Asthma Exacerbations
Keywords: Asthma; Asthma, Severe; Asthma Exacerbation; Emergency Treatment; Ketamine; Ketamine, Nebulized; Bronchodilator Agents; Randomized Controlled Trial; Peak Expiratory Flow Rate; Safety and Efficacy
MeSH Terms: conditions — Asthma | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: This is a prospective, double-blinded, randomized controlled trial using a parallel assignment model. Adult patients with moderate to severe asthma exacerbation are randomly assigned to one of two study arms:
  * Intervention group receiving nebulized ketamine (0.5 mg/kg) plus standard asthma care.
  * Control group receiving placebo nebulization (normal saline) plus standard asthma care.
  Participants remain in their assigned group throughout the study duration, and outcomes (e.g., peak expiratory flow rate, adverse events, symptom relief) are compared between groups to evaluate the efficacy and safety of nebulized ketamine.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study uses a double-blind design where all key parties are masked: participants, care providers (administering the nebulization), investigators (overseeing clinical care), and outcomes assessors (recording PEFR and symptom scores). Nebulized ketamine and placebo are prepared in identical-appearing formulations (5 mL clear solution in a nebulizer chamber) to maintain blinding. Randomization codes are securely stored and revealed only after data collection is complete. This design minimizes bias in treatment administration, symptom reporting, and outcome measurement
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nebulized ketamine (0.5 mg/kg) + standard care for moderate to severe asthma exacerbation (Experimental): Participants in the intervention arm will receive a single dose of nebulized ketamine at 0.5 mg/kg, diluted in normal saline to a total volume of 5ml, administered via a standard jet nebulizer. This will be given after standard asthma care, which includes salbutamol, ipratropium bromide, systemic corticosteroids (e.g., oral prednisolone or IV hydrocortisone), and supplemental oxygen as needed. The goal is to assess whether adding nebulized ketamine improves respiratory function, measured by peak expiratory flow rate (PEFR), compared to standard care alone. Participants will be monitored for 60 minutes after treatment for changes in PEFR, symptom relief, and any adverse effects. The intervention is non-invasive and administered in the emergency department for adult patients with moderate to severe asthma exacerbations.
  Interventions: Drug: Nebulized ketamine (0.5 mg/kg in normal saline to a total volume of 5ml) plus standard asthma excaerbationcare
- Placebo nebulization (normal saline) + standard care for moderate to severe asthma exacerbation (Placebo Comparator): Participants in the control arm will receive a placebo nebulization consisting of 5 mL of normal saline, administered via a standard jet nebulizer. This will be given in addition to standard asthma care, which includes salbutamol, ipratropium bromide, systemic corticosteroids (e.g., oral prednisolone or IV hydrocortisone), and supplemental oxygen as needed. The placebo is indistinguishable in appearance and administration method from the active treatment to maintain blinding. This arm is designed to evaluate the effects of standard care alone on peak expiratory flow rate (PEFR), symptom relief, and adverse events, and will be compared to the intervention group receiving nebulized ketamine. All participants will be monitored for 60 minutes following treatment in the emergency department setting.
  Interventions: Drug: Placebo nebulization (5 mL normal saline) plus standard asthma care

INTERVENTIONS:
Drug: Nebulized ketamine (0.5 mg/kg in normal saline to a total volume of 5ml) plus standard asthma excaerbationcare — **Intervention Description:** Nebulized ketamine is administered as a single dose of 0.5 mg/kg of ketamine hydrochloride diluted in 0.9% normal saline to a total volume of 5ml. The solution is delivered via a standard jet nebulizer over approximately 15-20minutes. This intervention is given once at the time of enrollment in the emergency department, in addition to standard asthma care. The ketamine used is in injectable solution form (typically 50 mg/mL concentration), drawn and diluted immediately prior to nebulization. Participants are monitored continuously for 60 minutes after administration to assess changes in peak expiratory flow rate (PEFR), symptom relief, and adverse events. The goal is to evaluate the bronchodilatory effect and safety of nebulized ketamine in adults with moderate to severe asthma exacerbation who present to the emergency department.
  Arms: Nebulized ketamine (0.5 mg/kg) + standard care for moderate to severe asthma exacerbation
Drug: Placebo nebulization (5 mL normal saline) plus standard asthma care — **Intervention Description (Control Group):** Participants in the control group will receive a single nebulized dose of 5 mL of 0.9% normal saline, delivered using a standard jet nebulizer over approximately 10-15 minutes. This placebo intervention is administered once at the time of enrollment in the emergency department, after standard asthma care. Standard care includes repeated doses of nebulized salbutamol and ipratropium, systemic corticosteroids (oral or intravenous), and supplemental oxygen as needed. The placebo solution is identical in appearance and volume to the active ketamine solution used in the intervention group to maintain blinding. All participants will be monitored for 60 minutes after nebulization to assess changes in peak expiratory flow rate (PEFR), symptom relief using a visual analog scale (VAS), and the occurrence of any adverse events.
  Arms: Placebo nebulization (normal saline) + standard care for moderate to severe asthma exacerbation

SUMMARY:
The goal of this clinical trial is to learn if nebulized ketamine helps treat moderate to severe asthma attacks in adults in the emergency department. It will also learn about the safety of ketamine when inhaled through a nebulizer.

The main questions it aims to answer are:

* Does nebulized ketamine improve breathing more than standard treatment alone?
* What side effects, if any, do participants experience after receiving nebulized ketamine?

Researchers will compare nebulized ketamine to a placebo (a saltwater mist with no medication) to see how well it works and how safe it is.

Participants will:

* Receive either nebulized ketamine or a placebo mist, along with standard asthma treatment
* Have their breathing checked before and after treatment using a peak flow meter
* Be monitored for 60 minutes and have their symptoms, vital signs, and any side effects recorded

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years or older presenting to the Emergency Department with a clinical diagnosis of moderate to severe asthma exacerbation based on SIGN (Scottish Intercollegiate Guidelines Network) criteria.
2. PEFR between 33% and 75% of predicted value or personal best, as measured using a peak flow meter.
3. Stable vital signs as deemed by the treating physician
4. Alert and oriented, able to understand the study purpose and provide informed consent.
5. Not requiring immediate advanced airway intervention, including intubation or emergency non-invasive ventilation.

Exclusion Criteria:

1. Known hypersensitivity or allergy to ketamine or any component of the nebulized solution.
2. History of psychosis, schizophrenia, or other severe uncontrolled psychiatric disorders.
3. Uncontrolled hypertension, defined as systolic BP > 180 mmHg or diastolic BP > 110 mmHg on two consecutive readings at least 5 minutes apart, despite initial ED management.
4. Hemodynamic instability, including persistent hypotension (SBP < 90 mmHg) or tachyarrhythmias requiring urgent treatment.
5. Significant chronic lung disease, including:

   * COPD with frequent exacerbations or baseline FEV₁ < 50% predicted
   * Interstitial lung disease (ILD)
   * Clinically significant bronchiectasis with baseline productive cough or infection
6. Pregnancy or currently breastfeeding.
7. Home BiPAP use or requirement for non-invasive ventilation (e.g., BiPAP/CPAP) during the ED visit (Note: isolated home CPAP for sleep apnea without daytime symptoms is acceptable).
8. Current intubation or imminent need for mechanical ventilation based on clinical judgment.
9. Severe cardiac disease, including decompensated heart failure, recent myocardial infarction (<6 weeks), or known severe valvular disease.
10. Any other medical, surgical, or psychiatric condition that in the opinion of the investigator would place the patient at undue risk from study participation or interfere with the interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Peak Expiratory Flow Rate (PEFR) from baseline to 60 minutes post-intervention | Baseline (0 minutes) and 60 minutes post-intervention
  PEFR will be measured using a peak flow meter at baseline (0 minutes) and at 60 minutes after administration of the intervention. The change in PEFR will be calculated to assess the intervention effect.

SECONDARY OUTCOMES:
Change in PEFR at 30 minutes | 30 minutes
• Incidence of adverse effects | 60 minutes
Incidence of intravenous magnesium sulfate administration | 60 minutes
  The proportion of participants who receive intravenous magnesium sulfate as part of escalation of care after 60 minutes post-intervention.
Incidence of ICU admission | 60 minutes
  The proportion of participants who require transfer to an intensive care unit (ICU) after 60 minutes post-intervention.
Incidence of endotracheal intubation | 60 minutes
  The proportion of participants who undergo endotracheal intubation after 60 minutes post-intervention due to clinical deterioration.
Incidence of non-invasive ventilation (BiPAP) initiation | 60 minutes
  The proportion of participants who require initiation of bilevel positive airway pressure (BiPAP) after 60 minutes post-intervention as part of escalation of care.
Disposition plan (discharged, admitted, or transferred) | 60 minutes
Length of stay (if admitted) | 60 minutes
Type of admission bed (e.g., ward vs. ICU) | 60 minutes
Change in dyspnea severity as measured by the Visual Analogue Scale (VAS) | 60 minutes
  Patient-reported breathlessness will be assessed using the Visual Analogue Scale (VAS), a 10-centimeter horizontal line ranging from 0 to 10. A score of 0 represents "no breathlessness," and a score of 10 represents "worst imaginable breathlessness." The change in VAS score from baseline to 60 minutes post-intervention will be recorded.